CLINICAL TRIAL: NCT07103070
Title: A Test of Efficacy and Foot Position Alteration in Patients Wearing Good Feet Arch Supports for the Treatment of Pain
Acronym: Good Feet
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Adam S. Landsman, DPM, PhD, Assistant Professor, Massachusetts General Hospital
Other Study IDs: 2022P000291
Record Dates: First submitted 2025-07-14; First posted 2025-08-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Plantar Fasciitis of Both Feet; Metatarsalgia; Morton Neuroma; Hallux Valgus Deformity; Low Back Pain; Knee Pain; Ankle Pain
Keywords: arch supports; heel pain; metatarsalgia; plantar fasciitis
MeSH Terms: conditions — Metatarsalgia; Morton Neuroma; Low Back Pain; Fasciitis, Plantar | interventions — Foot Orthoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inclusion 1. Men or women ≥ 18 and ≤ 65 years of age 2. The subject is able and willing to comply w: Subjects with foot pain who are able to wear arch supports.
  Interventions: Device: Arch supports

INTERVENTIONS:
Device: Arch supports — Set of 3 arch supports supplied by Good Feet

SUMMARY:
This study is a single armed prospective case series designed to evaluate the efficacy of treating common structural-related foot ailments (i.e. plantar fasciitis, metatarsalgia, and/or hallux valgus) with a high quality non-custom made arch support. It is believed that these conditions are the result of inadequate or poorly fitted arch supports resulting in a lack of structural correction in the foot while weight bearing. Over-the-counter insoles are believed to counteract the shortcomings in foot structure that result in these painful conditions. In this study, it is proposed that changes in foot morphology can be measured quantitatively using weight bearing CT Scan (Computerized Tomography) and X-rays of the subject with and without the arch supports. Subjects will also answer questions from a validated series of questionnaires pertaining to their foot condition and generalized health and activity level.

The study is a minimal risk study, with all subjects receiving the arch supports being investigated. There is no placebo offered. Initial evaluation of all subjects will include all imaging and measurements. Collection of subjective responses will occur after 4 weeks, 8 weeks, and 12 weeks of treatment.

DETAILED DESCRIPTION:
1. Background and Significance

   Foot orthoses are arch supports that can be worn in the shoes, and are designed to relieve pain by providing support to various areas of the foot to eliminate or reduce excessive mechanical forces. Most commonly, these devices are used as part of the treatment protocol for a variety of common foot ailments including painful plantar fasciitis and pronation. A variety of musculoskeletal pains have been shown to be reduced, and stability in ambulation can be improved by adding arch support to the shoes. Most importantly, previous studies have demonstrated that the structure of the foot can be altered, and with that the function of the foot, when orthoses are used.

   Previous studies have demonstrated multiple biomechanical and clinical benefits of using foot orthoses and arch supports. These devices have been shown to alter foot positioning and forefoot pressure during walking, reducing heel and forefoot pressures, decreasing impact forces, and improving comfort. Cadaveric studies confirm that orthoses enhance ankle and subtalar joint stability, correct abnormal rotations, improve arch alignment, and increase arch height under simulated load. Clinical studies involving military personnel found that wearing arch supports significantly reduced stress fracture incidence and improved comfort. Additionally, arch supports were associated with decreased lower back pain after prolonged use. Research also indicated that orthotic devices reduce tibial internal rotation, influencing the mechanical function of proximal structures like the ankle and leg. Furthermore, orthoses positively impacted foot deformities, pain (foot, knee, hip, and back), and balance, as demonstrated by radiographic and center-of-pressure analyses, indicating overall improvements in stability and symptomatic relief.

   The goal of the current study is to investigate the clinical and biomechanical effects of arch-support insoles in common foot pathologies including plantar fasciitis, and metatarsalgia.
2. Specific Aims and Objectives

   The objective of this study is to measure the structural changes that occur in the foot when wearing arch supports, and how these changes correlate with overall relief of common structural-related foot ailments; plantar fasciitis, metatarsalgia, and/or hallux valgus

   Specific Aim #1:

   Measure any changes that occur in the position and alignment of the foot bones relative to one another using weight bearing radiographs and weight bearing CT scans, with and without over-the-counter arch supports under the sole of the feet.

   Hypothesis: Arch supports (orthoses) will alter the positioning and alignment of the bones of the foot when standing. Any changes will be measurable in three dimensions, using both weight bearing CT scans and standard anterior-posterior and lateral radiographs.

   Specific Aim #2:

   Demonstrate if there is a correlation between symptomatic relief of painful foot conditions including plantar fasciitis and metatarsalgia pain using validated clinical scores and quality of life measures.

   Hypothesis: Painful foot conditions will improve when subjects wear over-the-counter arch supports on a regular basis, as demonstrated by validated subjective scoring.
3. General Description of Study Design

This study is a single armed prospective case series designed to evaluate the efficacy of treating common structural-related foot ailments (i.e. plantar fasciitis, metatarsalgia, and/or hallux valgus) with a high quality non-custom made arch support. It is believed that these conditions are the result of inadequate or poorly fitted arch supports resulting in a lack of structural correction in the foot while weight bearing. Over-the-counter insoles are believed to counteract the shortcomings in foot structure that result in these painful conditions. In this study, it is proposed that changes in foot morphology can be measured quantitatively using weight bearing CT Scan (Computerized Tomography) and X-rays of the subject with and without the arch supports. Subjects will also answer questions from a validated series of questionnaires pertaining to their foot condition and generalized health and activity level.

The study is a minimal risk study, with all subjects receiving the arch supports being investigated. There is no placebo offered. Initial evaluation of all subjects will include all imaging and measurements. Collection of subjective responses will occur after 4 weeks, 8 weeks, and 12 weeks of treatment.

Subject Recruitment:

Subjects will be recruited from the clinicians in the Division of Podiatry under the Department of Orthopaedics. Additionally, the sponsor, Good Feet Worldwide has a trade store the MGH service area, and will allow us to promote the study at their location with an advertisement poster. Potential subjects from the trade store will be referred to our clinics for screening and, when appropriate, recruited for the study.

Potential subjects will contact the principal investigator, Dr. Adam Landsman for preliminary screening and if they are able to satisfy the basic criteria, will be invited for formal screening. If qualified, they will be enrolled to begin the study. In order to avoid any undue pressure, all potential subjects who are patients of one of the Investigators will be given the option to do any or all of the following:

* Offer patients the opportunity to take home the Consent Form, and call back if they wish to participate
* Offer to connect the patient with other health care providers to discuss participation.

All study subjects will be screened and evaluated at the Foot and Ankle Clinic at MGH Waltham. Screenings and enrollments will take place on Tuesdays and Wednesdays, during dedicated research time.

The conditions being examined here are common among all races and genders, and enrollment is open to all. There have been limitations placed on subject age, as this age group is most likely to experience the conditions being studied.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 and ≤ 65 years of age
* Able and willing to comply with study procedures, and a signed and dated
* Diagnosed with symptomatic hallux valgus and/or plantar fasciitis and/or metatarsalgia
* Has had foot pain for at least 30 days
* Willing and able to utilize insole when walking for 90 days
* BMI ≤ 35
* Able to walk up to 0.5 miles without difficulty in a 24-hour period

Exclusion Criteria:

* Inability or unwillingness to comply with study procedures
* Gross asymmetry in feet, where shoe size differs by 2 or more full sizes between right and left foot
* Subject has had a CT performed within the last 30 days, for any body part.
* Prior partial or total amputation of a foot
* BMI > 35.
* Unilateral or bilateral foot deformity that would hinder the fitting of an over-the-counter arch support, such as active Charcot foot or Charcot with boney prominence
* Ulcers or open sores on either foot
* Currently wearing custom shoes or insoles.
* Currently ambulating with a cane, crutches, walker.
* Currently using any type of foot or ankle brace, and/or having used a brace in the last 30 days.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the clinicians in the Division of Podiatry under the Department of Orthopaedics. Additionally, the sponsor, Good Feet Worldwide has a trade store the MGH service area, and will allow us to promote the study at their location with an advertisement poster. Potential subjects from the trade store will be referred to our clinics for screening and, when appropriate, recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcome Measurement Information System (PROMIS)-Pain Intensity Score | 12 weeks
  Change in symptoms and relief of pain will be quantified based on subjective completion of validated questionnaires. Scoring is based on a 5-point scale, with higher scores indicating greater pain intensity. Raw scores are converted to T-scores, standardized to a mean of 50 (average for the general population) and a standard deviation of 10. Higher T-scores reflect more severe pain intensity.
Patient Reported Outcome Measurement Information System (PROMIS)-Pain Interference Score | 12 weeks
  PROMIS Pain Interference measures the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Respondents rate how much pain has interfered with their daily life over the past 7 days. Scoring uses a 5-point scale, with higher scores indicating greater interference. Raw scores are converted to T-scores (mean = 50, SD = 10); higher T-scores represent more significant pain interference.

SECONDARY OUTCOMES:
Change in foot morphology- Weightbearing X-ray | Baseline
  Foot alignment will be assessed using linear and angular measurements on anteroposterior and lateral views of plain radiographs. Images will be taken at baseline with and without insoles
Change in foot morphology- Weightbearing CT scans | Baseline
  Foot alignment will be assessed using 3D, linear, and angular measurements on CT scans. Images will be taken at baseline with and without insoles
Patient Reported Outcome Measurement Information System (PROMIS)-Global Health | 12 weeks
  PROMIS Global Health is a brief patient-reported outcome measure that assesses general physical, mental, and social health. It includes items covering overall health, quality of life, physical health, mental health, social roles, and symptom burden. Scoring is based on responses to a set of items (typically 4 or 10), each using a 5-point scale. Raw scores are converted to T-scores (mean = 50, SD = 10), with higher T-scores indicating better global health status.

CONTACTS AND LOCATIONS:
Overall Officials: Adam S Landsman, DPM, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
HIPPA compliance

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT07103070/Prot_SAP_000.pdf